CLINICAL TRIAL: NCT00856492
Title: A Randomized Phase II Trial of Weekly Nanoparticle Albumin Bound Paclitaxel (Nab-Paclitaxel) (NSC-736631) With or Without Bevacizumab, Either Preceded by or Followed by Q 2 Week Doxorubicin (A)and Cyclophosphamide (C) Plus Pegfilgrastim (PEG-G) as Neoadjuvant Therapy For Inflammatory and Locally Advanced HER-2/NEU Negative Breast Cancer
Brief Title: S0800, Nab-Paclitaxel, Doxorubicin, Cyclophosphamide, and Pegfilgrastim With or Without Bevacizumab in Treating Women With Inflammatory or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000636131; S0800 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; HER2-negative breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Bevacizumab; pegfilgrastim; Cyclophosphamide; Doxorubicin; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 and bevacizumab IV over 30- to 90-minutes on day 1 of weeks 1-12. Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 14, 16, 18, 20, 22, and 24.
  Interventions: Biological: bevacizumab; Biological: pegfilgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel albumin-stabilized nanoparticle formulation
- Arm 2 (Active Comparator): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 of weeks 1-12, and then receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 14, 16, 18, 20, 22, and 24.
  Interventions: Biological: pegfilgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel albumin-stabilized nanoparticle formulation
- Arm 3 (Active Comparator): Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 1, 3, 5, 7, 9, and 11, and then receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 of weeks 14-25.
  Interventions: Biological: pegfilgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel albumin-stabilized nanoparticle formulation

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Arms: Arm 1
Biological: pegfilgrastim — Given subcutaneously
Drug: cyclophosphamide — Given IV
Drug: doxorubicin hydrochloride — Given IV
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, doxorubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also may stop the growth of tumor cells by blocking blood flow to the tumor. Giving these treatments before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known which treatment regimen is more effective in treating women with breast cancer.

PURPOSE: This randomized phase II trial is studying paclitaxel albumin-stabilized nanoparticle formulation, doxorubicin, cyclophosphamide, and pegfilgrastim to compare how well they work when given with or without bevacizumab in treating women with inflammatory or locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the pathologic complete response rates in women with HER2/neu-negative inflammatory or locally advanced breast cancer treated with paclitaxel albumin-stabilized nanoparticle formulation, doxorubicin hydrochloride, cyclophosphamide, and pegfilgrastim with vs without bevacizumab.
* To compare the overall survival of patients treated with these regimens.
* To assess whether there is a correlation between bevacizumab and stratification factors (type of disease and hormone receptor status).
* To compare the toxicities of these regimens.
* To explore the molecular biomarkers related to the biology and outcome of inflammatory breast cancer.
* To explore potential molecular biomarkers that predict response to therapy and drug sensitivity.
* To evaluate biomarkers with respect to the sequence of paclitaxel albumin-stabilized nanoparticle formulation and doxorubicin hydrochloride/cyclophosphamide/pegfilgrastim administration in patients not receiving bevacizumab.
* To explore residual cancer burden and correlate it with outcome.
* To evaluate the time to treatment failure prior to surgery.
* To evaluate disease-free survival from the time of surgery in patients undergoing definitive surgery.

OUTLINE: This is a multicenter study. Patients are stratified according to type of disease (inflammatory vs locally advanced breast cancer) and hormone receptor status (positive [estrogen receptor (ER)+ and/or progesterone receptor (PgR)+] vs negative [ER- and PgR-]). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 and bevacizumab IV over 30- to 90-minutes on day 1 of weeks 1-12. Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 14, 16, 18, 20, 22, and 24.
* Arm II: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 of weeks 1-12. Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 14, 16, 18, 20, 22, and 24.
* Arm III: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 1, 3, 5, 7, 9, and 11. Patients then receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 of weeks 14-25.

In all arms, patients with stable or responding disease undergo surgery 3-6 weeks after completion of chemotherapy. Patients may then undergo radiotherapy 5 days a week for 6 weeks.

Serum, whole blood, and tissue samples are collected periodically for biomarker analysis, circulating endothelial cell analysis, and pharmacogenomic studies, respectively.

After completion of study treatment, patients are followed every 6 months for 1 year and then annually for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or pathologically confirmed breast cancer meeting one of the following criteria:

  * Locally advanced disease (stage IIIB disease, stage IIB/IIIA, or stage IIIC disease)
  * Inflammatory disease meeting the following two clinicopathologic criteria:

    * Diffuse erythema AND edema (peau d'orange) of the breast involving the majority of the skin of the breast, i.e., more than 50%
    * A biopsy demonstrating cancer either within the dermal lymphatics OR in the breast parenchyma itself
* HER2/neu-negative tumor as demonstrated by 0 or 1+ (weak or no staining) by DAKO, IHC, or equivalent test OR no gene amplification by FISH*

  * 2+ by DAKO or IHC allowed provided FISH* negative
* NOTE: *A negative FISH test ratio is < 1.8 or FISH HER2 gene copy < 4.0; if only a positive or negative result is available from the FISH test, a negative result is acceptable for study entry
* Hormone receptor status known

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Zubrod performance status 0-2
* Granulocyte count > 1,500/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin 9.0 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 mg/dL
* ALT and AST ≤ 3 times ULN
* Alkaline phosphatase ≤ 2.5 ULN (unless bone metastasis is present in the absence of liver metastasis)
* Urine protein:creatinine ratio ≤ 0.5 OR urine protein < 1,000 mg on 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to take oral medications (e.g., no uncontrolled nausea, vomiting, or diarrhea, lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome)
* QTc < 500 msec by EKG
* LVEF normal by MUGA or ECHO (for patients with hypertension or for patients > 60 years of age)
* NYHA class II cardiac function by baseline ECHO/MUGA (for patients who have received central thoracic radiotherapy that included the heart in the radiotherapy port, or for patients who have a history of class II heart failure but are asymptomatic on treatment are eligible)
* No history of stroke (cerebrovascular accident), transient ischemic attack, or cardiac event within the past 12 months, including any of the following:

  * Myocardial infarction (including severe/unstable angina)
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Pulmonary embolism
* No poorly controlled hypertension, defined as recurrent or persistent (≥ 24 hours) elevated blood pressure (i.e., systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg)
* No other malignancy within the past 5 years except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Peripheral neuropathy < grade 2

PRIOR CONCURRENT THERAPY:

* No prior tyrosine kinase inhibitors
* More than 5 years since prior chemotherapy, radiotherapy, or biologic therapy (e.g., trastuzumab or bevacizumab) for invasive breast cancer
* At least 7 days since prior hormonal therapy
* At least 7 days since prior and no concurrent strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole) or grapefruit juice
* No concurrent CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's wort)
* No other concurrent therapy for the treatment of breast cancer except for bisphosphonates
* No concurrent brachytherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (366):
- United States (365):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Breastlink Medical Group, Incorporated at Long Beach Memorial Medical Center, Long Beach, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Epic Care - Oakland, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center, Vallejo, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Singh and Arora Hematology Oncology, PC, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Great Lakes Cancer Institute - Lapeer Campus, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Erlanger Cancer Center at Erlanger Hospital - Baroness, Chattanooga, Tennessee
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Nab-Paclitaxel + Bevacizumab / AC+PEG-G)): Received intravenous (IV) administration of nabpaclitaxel 100 mg/m2 IV weekly for 12 weeks (nP x 12) with IV bevacizumab 10 mg/kg every 2 weeks (six doses), followed by IV doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 with pegfilgrastim 6 mg subcutaneously every 2 weeks for six cycles (ddAC x 6).
- Arm 2 (Nab-Paclitaxel / AC+PEG-G): Received nP x 12 without bevacizumab followed by ddAC x 6
- Arm 3 (AC+PEG-G / Nab-Paclitaxel): ddAC x 6 followed by nP x 12 without bevacizumab
Period: Overall Study
Arm/Group | Arm 1 (Nab-Paclitaxel + Bevacizumab / AC+PEG-G)) | Arm 2 (Nab-Paclitaxel / AC+PEG-G) | Arm 3 (AC+PEG-G / Nab-Paclitaxel)
Started | 99 | 63 | 53
Toxicity Eval (Fewer pts evaluable for toxicity vs arm totals b/c 2 pts on each arm did not receive any treatment) | 96 | 60 | 51
Completed | 98 | 62 | 51
Not Completed | 1 | 1 | 2
Not completed — Ineligible or withdrew consent | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 (Nab-Paclitaxel + Bevacizumab / AC+PEG-G): Received intravenous (IV) administration of nabpaclitaxel 100 mg/m2 IV weekly for 12 weeks (nP x 12) with IV bevacizumab 10 mg/kg every 2 weeks (six doses), followed by IV doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 with pegfilgrastim 6 mg subcutaneously every 2 weeks for six cycles (ddAC x 6).
- Arm 2 (Nab-Paclitaxel / AC+PEG-G)): Received nP x 12 followed by ddAC x 6 without bevacizumab
- Arm 3 (AC+PEG-G / Nab-Paclitaxel): Received ddAC x 6 first followed by nP x 12, without bevacizumab
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Nab-Paclitaxel + Bevacizumab / AC+PEG-G) | Arm 2 (Nab-Paclitaxel / AC+PEG-G)) | Arm 3 (AC+PEG-G / Nab-Paclitaxel) | Total
Number analyzed (Participants) | 98 | 62 | 51 | 211
Age, Continuous [Median (Full Range); unit: years] | 51.7 [22 to 71] | 49.7 [33 to 75] | 51.6 [31 to 66] | 51.5 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 62 | 51 | 211
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 70 | 44 | 40 | 154
  Race/Ethnicity: Black | 20 | 14 | 4 | 38
  Race/Ethnicity: Asian/Pacific Islander | 5 | 1 | 5 | 11
  Race/Ethnicity: Other/unknown | 3 | 3 | 2 | 8
Inflammatory Breast Cancer (IBC) or Non-IBC Locally Advanced Breast Cancer (LABC) [Count of Participants; unit: Participants]
  IBC | 10 | 7 | 7 | 24
  Non-IBC LABC | 88 | 55 | 44 | 187
Hormone receptor status [Count of Participants; unit: Participants]
  Positive: ER+ or PgR+ | 66 | 43 | 35 | 144
  Negative: ER- and PR- (TNBC) | 32 | 19 | 16 | 67
Breast cancer stage [Count of Participants; unit: Participants] — Measure Description: As per AJCC 6th ed, 2002:
  https://cancerstaging.org/references-tools/deskreferences/Documents/AJCC6thEdCancerStagingManualPart2.pdf Population: One subject missing Breast cancer stage information at baseline.
  Participants
    number analyzed (Participants) | 98 | 62 | 50 | 210
    IIB | 35 | 30 | 22 | 87
    IIIA | 32 | 16 | 14 | 62
    IIIB | 29 | 12 | 12 | 53
    IIIC | 2 | 4 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathological Complete Response Rate
Description: Pathologic complete response (pCR), commonly defined as the absence of residual invasive cancer in both the breast and axillary lymph nodes, has emerged as a surrogate endpoint for disease-free and overall survival, as the achievement of a pCR is associated with a favorable long-term prognosis in all breast cancer subtypes.
Time Frame: pre-study pathology vs. post-chemo surgery pathology (approx. 39-42 weeks post-randomization)
Population: Pre-specified analysis of Arm 1 vs. Arm 2/3 to compare effect of bevacizumab
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)): Received intravenous (IV) administration of nabpaclitaxel 100 mg/m2 IV weekly for 12 weeks (nP x 12) with IV bevacizumab 10 mg/kg every 2 weeks (six doses), followed by IV doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 with pegfilgrastim 6 mg subcutaneously every 2 weeks for six cycles (ddAC x 6).
- Arm 2/3 (Nab-Paclitaxel/AC+PEG-G)): Received nP x 12 followed by ddAC x 6, or received ddAC x 6 first followed by nP x 12, without bevacizumab
Arm/Group | Arm 1 (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) | Arm 2/3 (Nab-Paclitaxel/AC+PEG-G))
Number analyzed (Participants) | 98 | 113
Participants | 35 | 24
Statistical Analysis 1: Comparison: Arm 1 (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) vs Arm 2/3 (Nab-Paclitaxel/AC+PEG-G)); Test type: Superiority or Other; p = 0.019, Chi-squared

2. Secondary Outcome: Overall Survival
Description: Time from registration to death due to any cause
Time Frame: Disease assessed every 4 weeks while on treatment then every 6 months for one year then annually for four years from registration.
Population: Pre-specified analysis of Arm 1 vs. Arm 2/3 to compare effect of bevacizumab
Measure: Number; unit: deaths
Groups:
- Arm 2/3 (Nab-Paclitaxel/AC+PEG-G)): Arm II received nP x 12 followed by ddAC x 6, and those randomized to Arm III received ddAC x 6 first followed by nP x 12, both without bevacizumab
Arm/Group | Arm 1 (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) | Arm 2/3 (Nab-Paclitaxel/AC+PEG-G))
Number analyzed (Participants) | 98 | 113
deaths | 14 | 17
Statistical Analysis 1: Comparison: Arm 1 (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) vs Arm 2/3 (Nab-Paclitaxel/AC+PEG-G)); Test type: Superiority or Other; p = 0.64, Log Rank

3. Secondary Outcome: Event-free Survival
Description: Time from registration to first instance of any of the following events: progression prior to surgery, recurrence post-surgery or death from any cause.
Time Frame: Disease assessed every 4 weeks while on treatment then every 6 months for one year then annually for four years from registration or until recurrence
Population: Pre-specified analysis of Arm 1 vs. Arm 2/3 to compare effect of bevacizumab
Measure: Number; unit: participants
Arm/Group | Arm 1 (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) | Arm 2/3 (Nab-Paclitaxel/AC+PEG-G))
Number analyzed (Participants) | 98 | 113
participants | 20 | 24
Statistical Analysis 1: Comparison: Arm 1 (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) vs Arm 2/3 (Nab-Paclitaxel/AC+PEG-G)); Test type: Superiority or Other; p = 0.71, Log Rank

4. Secondary Outcome: Number of Adverse Events That Are Possibly, Probably or Definitely Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 28 weeks
Population: All participants receiving at least some protocol treatment
Measure: Number; unit: Participants
Groups:
- Arm I (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 and bevacizumab IV over 30- to 90-minutes on day 1 of weeks 1-12. Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 14, 16, 18, 20, 22, and 24.
- Arm II (Nab-Paclitaxel - AC+PEG-G): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 of weeks 1-12. Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 14, 16, 18, 20, 22, and 24.
- Arm III (AC+PEG-G - Nab-Paclitaxel): Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 2 of weeks 1, 3, 5, 7, 9, and 11. Patients then receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 of weeks 14-25.
Arm/Group | Arm I (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) | Arm II (Nab-Paclitaxel - AC+PEG-G) | Arm III (AC+PEG-G - Nab-Paclitaxel)
Number analyzed (Participants) | 96 | 60 | 51
Participants
  Abdominal pain | 2 | 0 | 0
  Adult respiratory distress syndrome | 1 | 0 | 0
  Alanine aminotransferase increased | 2 | 2 | 1
  Anemia | 13 | 6 | 13
  Anorectal infection | 2 | 0 | 0
  Anxiety | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1
  Blood and lymphatic system disorders - Other | 0 | 0 | 1
  Bone pain | 0 | 2 | 0
  CD4 lymphocytes decreased | 1 | 1 | 0
  Catheter related infection | 1 | 0 | 0
  Chest wall pain | 0 | 1 | 0
  Confusion | 1 | 0 | 0
  Conjunctivitis | 0 | 1 | 0
  Dehydration | 4 | 1 | 2
  Dental caries | 0 | 1 | 0
  Depression | 1 | 0 | 0
  Device related infection | 0 | 1 | 0
  Diarrhea | 3 | 1 | 1
  Dysphagia | 1 | 0 | 0
  Dyspnea | 3 | 0 | 1
  Ear pain | 1 | 0 | 0
  Edema limbs | 0 | 0 | 1
  Ejection fraction decreased | 1 | 0 | 1
  Enterocolitis | 0 | 0 | 1
  Enterocolitis infectious | 0 | 1 | 0
  Erythema multiforme | 1 | 0 | 0
  Facial nerve disorder | 1 | 0 | 0
  Facial pain | 0 | 1 | 0
  Fatigue | 7 | 7 | 4
  Febrile neutropenia | 10 | 5 | 3
  Gait disturbance | 0 | 1 | 0
  Gastrointestinal disorders - Other, specify | 1 | 0 | 0
  Generalized muscle weakness | 1 | 0 | 0
  Headache | 2 | 2 | 0
  Heart failure | 0 | 1 | 0
  Hypercalcemia | 0 | 1 | 0
  Hyperglycemia | 0 | 1 | 4
  Hypertension | 8 | 2 | 1
  Hypokalemia | 1 | 1 | 3
  Hyponatremia | 2 | 1 | 0
  Hypophosphatemia | 1 | 0 | 0
  Hypotension | 2 | 0 | 1
  Insomnia | 0 | 1 | 0
  Leukocytosis | 0 | 1 | 1
  Lung infection | 0 | 0 | 2
  Lymphocyte count decreased | 2 | 2 | 2
  Mucositis oral | 6 | 2 | 5
  Myalgia | 0 | 1 | 0
  Nasal congestion | 0 | 1 | 1
  Nausea | 6 | 6 | 4
  Neutrophil count decreased | 36 | 10 | 16
  Non-cardiac chest pain | 0 | 1 | 0
  Oral pain | 0 | 1 | 0
  Otitis externa | 1 | 0 | 0
  Pain | 2 | 2 | 0
  Pain in extremity | 0 | 1 | 1
  Palmar-plantar erythrodysesthesia syndrome | 1 | 0 | 2
  Periorbital infection | 1 | 0 | 0
  Peripheral motor neuropathy | 0 | 1 | 0
  Peripheral sensory neuropathy | 5 | 5 | 2
  Platelet count decreased | 6 | 3 | 0
  Pneumonitis | 2 | 0 | 2
  Proctitis | 1 | 0 | 0
  Proteinuria | 0 | 1 | 0
  Rash maculo-papular | 0 | 1 | 0
  Rectal pain | 0 | 1 | 0
  Renal and urinary disorders - Other, specify | 1 | 0 | 0
  Respiratory failure | 1 | 1 | 0
  Sepsis | 2 | 1 | 0
  Skin and subcutaneous tissue disorders - Other | 1 | 0 | 0
  Skin infection | 2 | 2 | 1
  Suicide attempt | 1 | 0 | 0
  Syncope | 1 | 0 | 1
  Thromboembolic event | 1 | 2 | 0
  Tooth infection | 0 | 1 | 1
  Urinary tract infection | 1 | 1 | 1
  Vomiting | 9 | 3 | 2
  Vulval infection | 1 | 0 | 0
  Weight gain | 1 | 0 | 0
  Weight loss | 0 | 0 | 1
  White blood cell decreased | 15 | 5 | 12

ADVERSE EVENTS:
Time Frame: Up to 25 weeks
Arm/Group | Arm I (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) | Arm II (Nab-Paclitaxel - AC+PEG-G) | Arm III (AC+PEG-G - Nab-Paclitaxel)
Serious Adverse Events (participants affected / at risk) | 22/96 | 3/60 | 3/51
Other Adverse Events (participants affected / at risk) | 92/96 | 58/60 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) (N=96) | Arm II (Nab-Paclitaxel - AC+PEG-G) (N=60) | Arm III (AC+PEG-G - Nab-Paclitaxel) (N=51)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0
Heart failure (Cardiac disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1
Death NOS (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 0
Skin infection (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Investigations-Other (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 5 | 0 | 2
Platelet count decreased (Investigations) | 1 | 1 | 0
Weight gain (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 4 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Thromboembolic event (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nab-Paclitaxel + Bevacizumab - AC+PEG-G)) (N=96) | Arm II (Nab-Paclitaxel - AC+PEG-G) (N=60) | Arm III (AC+PEG-G - Nab-Paclitaxel) (N=51)
Anemia (Blood and lymphatic system disorders) | 73 | 43 | 48
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 3
Sinus tachycardia (Cardiac disorders) | 5 | 1 | 2
Ear pain (Ear and labyrinth disorders) | 4 | 1 | 4
Blurred vision (Eye disorders) | 6 | 8 | 5
Conjunctivitis (Eye disorders) | 2 | 1 | 4
Dry eye (Eye disorders) | 3 | 2 | 3
Eye disorders-Other (Eye disorders) | 5 | 4 | 2
Watering eyes (Eye disorders) | 20 | 7 | 11
Abdominal pain (Gastrointestinal disorders) | 13 | 7 | 8
Anal pain (Gastrointestinal disorders) | 4 | 3 | 0
Bloating (Gastrointestinal disorders) | 4 | 1 | 4
Constipation (Gastrointestinal disorders) | 52 | 24 | 26
Diarrhea (Gastrointestinal disorders) | 46 | 31 | 27
Dry mouth (Gastrointestinal disorders) | 5 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 17 | 7 | 15
Dysphagia (Gastrointestinal disorders) | 9 | 2 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 4 | 5
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 6 | 2 | 2
Hemorrhoids (Gastrointestinal disorders) | 6 | 1 | 4
Mucositis oral (Gastrointestinal disorders) | 42 | 26 | 29
Nausea (Gastrointestinal disorders) | 73 | 49 | 41
Oral pain (Gastrointestinal disorders) | 5 | 1 | 3
Rectal hemorrhage (Gastrointestinal disorders) | 6 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 3 | 1
Vomiting (Gastrointestinal disorders) | 35 | 32 | 28
Chills (General disorders) | 14 | 7 | 8
Edema limbs (General disorders) | 8 | 12 | 9
Fatigue (General disorders) | 85 | 50 | 45
Fever (General disorders) | 12 | 7 | 12
Flu like symptoms (General disorders) | 4 | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 4 | 2
Pain (General disorders) | 34 | 23 | 10
Bronchial infection (Infections and infestations) | 1 | 1 | 3
Infections and infestations-Other (Infections and infestations) | 3 | 2 | 4
Lung infection (Infections and infestations) | 2 | 0 | 3
Nail infection (Infections and infestations) | 14 | 2 | 2
Sinusitis (Infections and infestations) | 6 | 2 | 1
Skin infection (Infections and infestations) | 10 | 4 | 7
Tooth infection (Infections and infestations) | 2 | 4 | 2
Upper respiratory infection (Infections and infestations) | 8 | 3 | 8
Urinary tract infection (Infections and infestations) | 7 | 6 | 4
Alanine aminotransferase increased (Investigations) | 31 | 18 | 16
Alkaline phosphatase increased (Investigations) | 20 | 8 | 16
Aspartate aminotransferase increased (Investigations) | 25 | 17 | 19
CD4 lymphocytes decreased (Investigations) | 1 | 1 | 3
Creatinine increased (Investigations) | 8 | 2 | 2
Investigations-Other (Investigations) | 10 | 2 | 3
Lymphocyte count decreased (Investigations) | 6 | 3 | 8
Neutrophil count decreased (Investigations) | 58 | 24 | 26
Platelet count decreased (Investigations) | 21 | 11 | 13
Weight loss (Investigations) | 27 | 6 | 13
White blood cell decreased (Investigations) | 48 | 22 | 29
Anorexia (Metabolism and nutrition disorders) | 35 | 19 | 20
Dehydration (Metabolism and nutrition disorders) | 8 | 5 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 32 | 14 | 19
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 7 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 21 | 6 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 22 | 11 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 14 | 4 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 12 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 4 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 12 | 13
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 8 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 9 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 10 | 8
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 3
Dizziness (Nervous system disorders) | 23 | 12 | 16
Dysgeusia (Nervous system disorders) | 35 | 11 | 9
Headache (Nervous system disorders) | 45 | 26 | 19
Memory impairment (Nervous system disorders) | 4 | 3 | 1
Paresthesia (Nervous system disorders) | 3 | 4 | 1
Peripheral motor neuropathy (Nervous system disorders) | 4 | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 69 | 40 | 30
Anxiety (Psychiatric disorders) | 15 | 10 | 7
Depression (Psychiatric disorders) | 17 | 9 | 9
Insomnia (Psychiatric disorders) | 33 | 15 | 10
Proteinuria (Renal and urinary disorders) | 7 | 2 | 1
Urinary frequency (Renal and urinary disorders) | 4 | 0 | 3
Urinary tract pain (Renal and urinary disorders) | 5 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 16 | 10 | 6
Irregular menstruation (Reproductive system and breast disorders) | 3 | 4 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 3 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 17 | 4 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 14 | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 36 | 19 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 43 | 5 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 | 9 | 6
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 16 | 5 | 5
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 56 | 37 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 7 | 10
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 | 3 | 4
Nail discoloration (Skin and subcutaneous tissue disorders) | 30 | 15 | 19
Nail loss (Skin and subcutaneous tissue disorders) | 13 | 5 | 8
Nail ridging (Skin and subcutaneous tissue disorders) | 13 | 5 | 6
Pain of skin (Skin and subcutaneous tissue disorders) | 7 | 2 | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 10 | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 13 | 7 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 37 | 10 | 10
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 12 | 5 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 14 | 5 | 3
Flushing (Vascular disorders) | 5 | 1 | 1
Hot flashes (Vascular disorders) | 20 | 11 | 13
Hypertension (Vascular disorders) | 36 | 10 | 5
Hypotension (Vascular disorders) | 12 | 5 | 4
Thromboembolic event (Vascular disorders) | 5 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less